CLINICAL TRIAL: NCT01939158
Title: A PHASE III, RANDOMISED, OPEN, CONTROLLED, MULTICENTRE, PRIMARY VACCINATION STUDY TO EVALUATE THE IMMUNOGENICITY AND PERSISTENCE OF 1 AND 2 DOSES OF MENINGOCOCCAL CONJUGATE VACCINE MENACWY-TT IN TODDLERS (AFTER 1 MONTH AND UP TO 5 YEARS) AND TO DEMONSTRATE NON-INFERIORITY OF CO-ADMINISTRATION OF MENACWY-TT AND 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE PREVENAR 13(REGISTERED) VERSUS SEPARATE ADMINISTRATION OF THE 2 VACCINES
Brief Title: Immunogenicity and Safety Study of 1 and 2 Doses of GlaxoSmithKline (GSK) Biologicals' Meningococcal Vaccine MenACWY-TT (GSK134612) in Toddlers, Persistence up to 5 Years After Vaccination and Co-administration With Pfizer's Prevenar 13™Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MENACWY-TT-104; C0921003 (Other: Alias Study Number); 2013-001083-28 (EudraCT Number); 116892 (Other: Alias Study Number)
Record Dates: First submitted 2013-08-29; First posted 2013-09-11 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Infections, Meningococcal
Keywords: Co-administration; Safety; Persistence; Immunogenicity; Prevenar 13; Meningococcal vaccine; Toddlers; 5 years
MeSH Terms: conditions — Meningococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ACWY1d group (Experimental): Subjects will receive 1 dose of the MenACWY-TT vaccine
  Interventions: Biological: Meningococcal vaccine GSK134612
- ACWY2d group (Experimental): Subjects will receive 2 doses of the MenACWY-TT vaccine 2 months apart
  Interventions: Biological: Meningococcal vaccine GSK134612
- Co-ad group (Experimental): Subjects will receive 1 dose of the MenACWY-TT vaccine co-administered with Prevenar 13™
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Prevenar 13™
- PCV-13 group (Active Comparator): Subjects will receive 1 dose of Prevenar 13™ and 1 dose of the MenACWY-TT vaccine 2 months later
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Prevenar 13™

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — 1 or 2 doses administered intramuscularly in the left anterolateral thigh or deltoid region
Biological: Prevenar 13™ — 1 dose administered intramuscularly in the right anterolateral thigh or deltoid region
  Arms: Co-ad group; PCV-13 group

SUMMARY:
The purpose of this study is to compare the immediate and long term (up to 5 years) immunogenicity and safety of GSK Biologicals' MenACWY-TT vaccine when given as a single dose or as 2 doses to toddlers aged 12 to 14 months. Also, this study will also assess if co-administration of GSK Biologicals' MenACWY-TT with the booster dose of Pfizer's Prevenar 13 adversely impacts the immunogenicity of either of the vaccines.

DETAILED DESCRIPTION:
The Medicines Control Council (MCC) authorities requested that subjects be screened for HIV testing prior to study enrolment in South Africa to ensure that only HIV negative participants are enrolled. As such, HIV rapid test was added at Visit 1 only for subjects in South Africa. Subjects previously screened HIV positive will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 14 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Vaccination records showing the completion of the full primary vaccination schedule with Prevenar 13 and Diphtheria, Tetanus and Pertussis (DTP) containing vaccine according to local recommendations at least 5 months before the study entry.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after the dose of vaccines, with the exception of a licensed inactivated influenza vaccine. Measles, Mumps Rubella (MMR) vaccine or Measles Mumps Rubella and Varicella (MMRV) vaccine can be co-administered with MenACWY-TT and/or Prevenar 13. A DTPa containing vaccine can be administered after the last blood sampling (at Visit 2 or 4 depending on the group).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against Neisseria meningitidis.
* Previous booster vaccination against Streptococcus pneumoniae.
* Previous booster vaccination against Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination (no laboratory testing required)*

  * Note: With the exception of HIV rapid testing which will be done for subjects in South Africa.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity, including to diphtheria toxoid, likely to be exacerbated by any component of the vaccines.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures, including Guillain-Barré syndrome (GBS). History of a simple, single febrile seizure is permitted.
* Acute disease and/or fever at the time of enrollment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 12 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 803 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- Australia (5):
  - Canberra Hospital, Garran, Australian Capital Territory
  - The Childrens Hospital at Westmead, Westmead, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Vaccine and Immunization Research Group, Melbourne, Victoria
  - Vaccine Trials Group, Telethon Kids Institute, Perth Children's Hospital, Nedlands, Western Australia
- Canada (5):
  - The Clinical Research Unit; Children's Hospital Research Institute of Manitoba [CHRIM], Winnipeg, Manitoba
  - Canadian Center for Vaccinology - IWK Health Centre, Halifax, Nova Scotia
  - Medicor Research Inc., Greater Sudbury, Ontario
  - Dr. Allen Greenspoon Medicine Professional Corporation, Hamilton, Ontario
  - CHU de Quebec-Universite Laval, Québec, Quebec
- Czechia (29):
  - Medicentrum 6 s.r.o, Prague, Vokovice
  - Ordinace praktickeho lekare pro deti a dorost, Benešov
  - Ordinace praktickeho lekare pro deti a dorost, Boletice nad Labem
  - Ordinace praktickeho lekare pro deti a dorost, Brandýs nad Labem
  - Ordinace praktickeho lekare pro deti a dorost, Chrastava
  - Ordinace praktickeho lekare pro deti a dorost, Chrudim
  - Ordinace praktickeho lekare pro deti a dorost, Čáslav
  - Krajska zdravotni, a.s., Nemocnice Decin, Děčín
  - Ordinace praktickeho lekare pro deti a dorost, Domažlice
  - Ordinace praktickeho lekare pro deti a dorost, Holice
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Hrádek nad Nisou
  - Ordinace praktickeho lekare pro deti a dorost, Hronov
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Ordinace Praktickeho Lekare Pro Deti A Dorost, Kladno
  - Ordinace praktickeho lekare pro deti a dorost, Krupka
  - Ordinace praktickeho lekare pro deti a dorost, Liberec
  - Ordinace praktickeho lekare pro deti a dorost, Mělník
  - Oblastni nemocnice Nachod, Náchod
  - Ordinace praktickeho lekare pro deti a dorost, Neveklov
  - Ordinace praktickeho lekare pro deti a dorost, Nový Jičín
  - Ordinace Praktickeho Lekare pro deti a dorost, Odolena Voda
  - Ordinace praktickeho lekare pro deti a dorost, Ostrov
  - Ordinace praktickeho lekare pro deti a dorost, Pardubice
  - Nemocnice Pardubice, Pardubice
  - Ordinace praktickeho lekare pro deti a dorost, Prague
  - Ordinace praktickeho lekare pro deti a dorost, Smiřice
  - Ordinace Praktickeho Lekare pro deti a dorost, Trutnov
  - Ordinace praktickeho lekare pro deti a dorost, Týnec nad Sázavou
- Panama (4):
  - Centro Pediatrico America, Consultorios America, Panama City
  - CEVAXIN Plaza Carolina, Panama City
  - Consultorios America Via Espana, Panama City
  - ULAPS Guadalupe, Panama City
- South Africa (2):
  - Chris Hani Baragwanath Academic Hospital, Soweto, Gauteng
  - Setshaba Clinical Research, Gauteng
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Medicine, Ankara, Sihhiye
  - Ege University Hospital Medical Faculty, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cutland CL, Peyrani P, Webber C, Newton R, Cutler M, Perez JL. A phase 3, randomized, controlled, open-label study to evaluate the persistence up to 5 years of 1 or 2 doses of meningococcal conjugate vaccine MenACWY-TT given with or without 13-valent pneumococcal conjugate vaccine in 12-14-month-old children. Vaccine. 2023 Jan 27;41(5):1153-1160. doi: 10.1016/j.vaccine.2022.11.048. Epub 2023 Jan 6. PMID 36621408
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=MENACWY-TT-104&StudyName=A+Phase+Iii%2C+Randomised%2C+Open%2C+Controlled%2C+Multicentre%2C+Primary+Vaccination+Study+To+Evaluate+The+Immunogenicity+And+Persistence+Of+1+And+2+Doses+Of+Meningococcal+Conjugate+Vaccine+Menacwy-tt+In+Toddlers+%28after+1+Month+And+Up+To+5+Years%29+And+To+Demonstrate+Non-inferiority+Of+Co-administration+Of+Menacwy-tt+And+13-valent+Pneumococcal+Conjugate+Vaccine+Prevenar+13%28registered%29+Versus+Separate+Administration+Of+The+2+Vaccines

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from 2 October 2013 to 5 December 2019.
Pre-assignment Details: A total of 803 participants were enrolled and were randomized in 1:1:1:1 ratio to either ACWY1d, ACWY2d, Co-ad and PCV13 groups.
Groups:
- ACWY1d Group: Participants received single dose of meningococcal polysaccharide groups A, C, W-135, and Y tetanus toxoid conjugate (MenACWY-TT) vaccine administered intramuscularly at Month 0.
- ACWY2d Group: Participants received two doses of MenACWY-TT vaccine administered intramuscularly at Month 0 and Month 2.
- Co-ad Group: Participants received single dose of MenACWY-TT vaccine and single dose of Prevnar 13 administered intramuscularly at Month 0.
- PCV13 Group: Participants received single dose of Prevnar 13 at Month 0 and single dose of MenACWY-TT administered intramuscularly at Month 2.
Period: Overall Study
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Started | 203 | 198 | 201 | 201
Vaccinated | 203 | 197 | 201 | 201
Completed | 156 | 146 | 160 | 157
Not Completed | 47 | 52 | 41 | 44
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 22 | 25 | 15 | 17
Not completed — Migrated/moved from study area | 5 | 7 | 3 | 6
Not completed — Lost to Follow-up | 18 | 17 | 17 | 17
Not completed — Death | 0 | 0 | 1 | 1
Not completed — No longer meets eligibility criteria | 0 | 0 | 1 | 0
Not completed — Other | 1 | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on participants, who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group | Total
Number analyzed (Participants) | 203 | 197 | 201 | 201 | 802
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.8 (0.9) | 12.8 (0.9) | 12.8 (0.9) | 12.7 (0.9) | 12.8 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 85 | 98 | 98 | 375
  Male | 109 | 112 | 103 | 103 | 427
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 7 | 8 | 31
  Not Hispanic or Latino | 195 | 189 | 194 | 193 | 771
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 3 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 33 | 33 | 31 | 30 | 127
  White | 135 | 127 | 137 | 134 | 533
  More than one race | 34 | 34 | 29 | 33 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Rabbit Complement Antibody (rSBA) Titers >=1:8 at 1 Month After Administration of 1 Dose of MenACWY-TT in the ACWY1d, ACWY2d and Co-ad Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 against each serogroup at 1 month after administration of MenACWY-TT are reported. According-to-protocol (ATP) cohort for persistence Year 1 population included all participants who met all eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present with a medical condition or received product leading to exclusion or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 1)
Population: Analyzed on ATP cohort for persistence Year 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for PCV13 reporting group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group
Number analyzed (Participants) | 180 | 158 | 178
percentage of participants
  rSBA-MenA | 97.8 [94.4 to 99.4] | 96.8 [92.8 to 99.0] | 94.9 [90.6 to 97.7]
  rSBA-MenC: number analyzed (Participants) | 179 | 157 | 176
  rSBA-MenC | 95.0 [90.7 to 97.7] | 95.5 [91.0 to 98.2] | 96.0 [92.0 to 98.4]
  rSBA-MenW-135: number analyzed (Participants) | 180 | 158 | 177
  rSBA-MenW-135 | 95.0 [90.7 to 97.7] | 94.9 [90.3 to 97.8] | 93.2 [88.5 to 96.4]
  rSBA-MenY: number analyzed (Participants) | 180 | 157 | 177
  rSBA-MenY | 92.8 [88.0 to 96.1] | 93.6 [88.6 to 96.9] | 89.8 [84.4 to 93.9]

2. Primary Outcome: Percentage of Participants With rSBA Titers >=1:8 at 1 Month After Administration of 2 Doses of MenACWY-TT in the ACWY2d Group
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 against each serogroup at 1 month after administration of 2 doses of MenACWY-TT are reported. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 2nd dose of MenACWY-TT (i.e. at Month 3)
Population: Analyzed on ATP cohort for persistence Year 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for ACWY1d, Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY2d Group
Number analyzed (Participants) | 150
percentage of participants
  rSBA-MenA | 98.0 [94.3 to 99.6]
  rSBA-MenC | 98.7 [95.3 to 99.8]
  rSBA-MenW-135 | 100.0 [97.6 to 100.0]
  rSBA-MenY | 99.3 [96.3 to 100.0]

3. Primary Outcome: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 at Year 1 in the ACWY1d and ACWY2d Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 and >=1:128 against each serogroup at Year 1 after administration of MenACWY-TT are reported. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 1
Population: Analyzed on ATP cohort for persistence Year 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 167 | 143
percentage of participants
  rSBA-MenA: >=1:8 | 63.5 [55.7 to 70.8] | 70.6 [62.4 to 77.9]
  rSBA-MenC: >=1:8 | 49.1 [41.3 to 56.9] | 55.2 [46.7 to 63.6]
  rSBA-MenW-135: >=1:8 | 65.3 [57.5 to 72.5] | 77.6 [69.9 to 84.2]
  rSBA-MenY: >=1:8 | 73.1 [65.7 to 79.6] | 79.7 [72.2 to 86.0]
  rSBA-MenA: >=1:128 | 44.9 [37.2 to 52.8] | 50.3 [41.9 to 58.8]
  rSBA-MenC: >=1:128 | 21.0 [15.1 to 27.9] | 27.3 [20.2 to 35.3]
  rSBA-MenW-135: >=1:128 | 46.7 [39.0 to 54.6] | 60.1 [51.6 to 68.2]
  rSBA-MenY: >=1:128 | 52.1 [44.2 to 59.9] | 60.8 [52.3 to 68.9]

4. Primary Outcome: Geometric Mean Titers (GMTs) With rSBA for Each of the 4 Serogroups Following Vaccination at Year 1 in the ACWY1d and ACWY2d Groups
Description: Geometric mean titers of antibodies against each serogroup were assessed using rSBA. Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). rSBA titers are expressed as 1/dilution. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 167 | 143
titers (1/dilution)
  rSBA-MenA | 62.7 [42.6 to 92.2] | 76.6 [50.7 to 115.7]
  rSBA-MenC | 16.2 [12.4 to 21.1] | 21.2 [15.6 to 28.9]
  rSBA-MenW-135 | 57.2 [39.9 to 82.0] | 123.1 [82.7 to 183.4]
  rSBA-MenY | 76.8 [54.2 to 109.0] | 112.3 [77.5 to 162.8]

5. Primary Outcome: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 at Year 3 in the ACWY1d and ACWY2d Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 and >=1:128 against each serogroup at Year 3 after administration of MenACWY-TT are reported. ATP cohort for persistence Year 3 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 3
Population: Analyzed on ATP cohort for persistence Year 3 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 147 | 121
percentage of participants
  rSBA-MenA: >=1:8 | 46.9 [38.7 to 55.3] | 54.5 [45.2 to 63.6]
  rSBA-MenC: >=1:8 | 35.4 [27.7 to 43.7] | 33.9 [25.5 to 43.0]
  rSBA-MenW-135: >=1:8 | 59.2 [50.8 to 67.2] | 72.7 [63.9 to 80.4]
  rSBA-MenY: >=1:8 | 61.9 [53.5 to 69.8] | 68.6 [59.5 to 76.7]
  rSBA-MenA: >=1:128 | 34.0 [26.4 to 42.3] | 31.4 [23.3 to 40.5]
  rSBA-MenC: >=1:128 | 9.5 [5.3 to 15.5] | 15.7 [9.7 to 23.4]
  rSBA-MenW-135: >=1:128 | 42.9 [34.7 to 51.3] | 52.9 [43.6 to 62.0]
  rSBA-MenY: >=1:128 | 49.0 [40.7 to 57.3] | 53.7 [44.4 to 62.8]

6. Primary Outcome: Geometric Mean Titers (GMTs) With rSBA for Each of the 4 Serogroups Following Vaccination at Year 3 in the ACWY1d and ACWY2d Groups
Description: Geometric mean titers of antibodies against each serogroup were assessed using rSBA. Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). rSBA titers are expressed as 1/dilution. ATP cohort for persistence Year 3 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 3
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 147 | 121
titers (1/dilution)
  rSBA-MenA | 29.7 [19.8 to 44.5] | 28.5 [18.7 to 43.6]
  rSBA-MenC | 9.8 [7.6 to 12.7] | 11.5 [8.4 to 15.8]
  rSBA-MenW-135 | 42.5 [29.2 to 61.8] | 92.9 [59.9 to 143.9]
  rSBA-MenY | 58.0 [39.1 to 86.0] | 75.1 [48.7 to 115.9]

7. Primary Outcome: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 at Year 5 in the ACWY1d and ACWY2d Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 and >=1:128 against each serogroup at Year 5 after administration of MenACWY-TT are reported. ATP cohort for persistence Year 5 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 5
Population: Analyzed on ATP cohort for persistence Year 5 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 133 | 117
percentage of participants
  rSBA-MenA: >=1:8 | 58.6 [49.8 to 67.1] | 65.8 [56.5 to 74.3]
  rSBA-MenC: >=1:8: number analyzed (Participants) | 132 | 116
  rSBA-MenC: >=1:8 | 20.5 [13.9 to 28.3] | 28.4 [20.5 to 37.6]
  rSBA-MenW-135: >=1:8 | 44.4 [35.8 to 53.2] | 50.4 [41.0 to 59.8]
  rSBA-MenY: >=1:8 | 47.4 [38.7 to 56.2] | 58.1 [48.6 to 67.2]
  rSBA-MenA: >=1:128 | 43.6 [35.0 to 52.5] | 53.0 [43.5 to 62.3]
  rSBA-MenC: >=1:128: number analyzed (Participants) | 132 | 116
  rSBA-MenC: >=1:128 | 6.1 [2.7 to 11.6] | 10.3 [5.5 to 17.4]
  rSBA-MenW-135: >=1:128 | 32.3 [24.5 to 41.0] | 39.3 [30.4 to 48.8]
  rSBA-MenY: >=1:128 | 39.8 [31.5 to 48.7] | 52.1 [42.7 to 61.5]

8. Primary Outcome: Geometric Mean Titers (GMTs) With rSBA for Each of the 4 Serogroups Following Vaccination at Year 5 in the ACWY1d and ACWY2d Groups
Description: Geometric mean titers of antibodies against each serogroup were assessed using rSBA. Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). rSBA titers are expressed as 1/dilution. ATP cohort for persistence Year 5 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 5
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 133 | 117
titers (1/dilution)
  rSBA-MenA | 46.8 [30.7 to 71.5] | 69.9 [44.7 to 109.3]
  rSBA-MenC: number analyzed (Participants) | 132 | 116
  rSBA-MenC | 6.6 [5.3 to 8.2] | 8.5 [6.4 to 11.2]
  rSBA-MenW-135 | 25.0 [16.7 to 37.6] | 37.1 [23.3 to 59.0]
  rSBA-MenY | 36.5 [23.6 to 56.2] | 55.8 [35.7 to 87.5]

9. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies for Each of the Anti-pneumococcal Serotypes at 1 Month After Administration of Prevnar 13 in the Co-ad and PCV-13 Groups
Description: GMCs for anti-pneumococcal antibodies (anti-1, anti-3, anti-4, anti-5, anti-6A, anti-6B, anti-7F, anti-9V, anti-14, anti-18C, anti-19A, anti-19F and anti-23F) were measured in microgram per milliliter (mcg/mL). ATP cohort for immunogenicity post dose 1 included all evaluable participants who met eligibility criteria, complied with the procedures defined in the protocol and with no elimination criteria during the study from the ATP cohort for safety, received all study vaccines at Month 0, had assay results available for antibodies against at least one study vaccine antigen component at Visit 2 (Month 1), and had available blood sample at Visit 2 (Month 1) for PCV13 group.
Time Frame: 1 month after administration of Prevnar 13 (i.e. at Month 1)
Population: Analyzed on ATP cohort for immunogenicity post dose 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for ACWY1d and ACWY2d reporting groups.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 163 | 172
mcg/mL
  anti-1: number analyzed (Participants) | 162 | 171
  anti-1 | 2.94 [2.56 to 3.36] | 2.62 [2.27 to 3.01]
  anti-3: number analyzed (Participants) | 151 | 162
  anti-3 | 0.80 [0.69 to 0.91] | 0.71 [0.62 to 0.81]
  anti-4 | 2.46 [2.14 to 2.83] | 1.96 [1.69 to 2.26]
  anti-5 | 2.09 [1.84 to 2.37] | 1.67 [1.46 to 1.91]
  anti-6A: number analyzed (Participants) | 163 | 171
  anti-6A | 8.59 [7.50 to 9.85] | 7.28 [6.33 to 8.37]
  anti-6B: number analyzed (Participants) | 161 | 171
  anti-6B | 7.36 [6.33 to 8.55] | 6.68 [5.70 to 7.83]
  anti-7F | 5.14 [4.49 to 5.88] | 4.81 [4.23 to 5.47]
  anti-9V | 2.03 [1.78 to 2.30] | 1.79 [1.59 to 2.03]
  anti-14: number analyzed (Participants) | 161 | 172
  anti-14 | 13.1 [11.38 to 15.07] | 11.94 [10.43 to 13.66]
  anti-18C | 2.53 [2.19 to 2.92] | 2.13 [1.84 to 2.47]
  anti-19A: number analyzed (Participants) | 162 | 170
  anti-19A | 9.60 [8.41 to 10.97] | 8.62 [7.53 to 9.87]
  anti-19F: number analyzed (Participants) | 162 | 172
  anti-19F | 8.40 [7.33 to 9.62] | 7.98 [6.96 to 9.15]
  anti-23F: number analyzed (Participants) | 161 | 169
  anti-23F | 5.33 [4.57 to 6.21] | 4.47 [3.83 to 5.23]

10. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titers >=1:4 and >=1:8 at 1 Month After Administration of 1 Dose of MenACWY-TT in the ACWY1d and ACWY2d Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with hSBA titers >=1:4 and >=1:8 against each serogroup at 1 month after administration of MenACWY-TT are reported. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 1)
Population: Analyzed on ATP cohort for persistence Year 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 78 | 70
percentage of participants
  hSBA-MenA: >=1:4: number analyzed (Participants) | 74 | 66
  hSBA-MenA: >=1:4 | 95.9 [88.6 to 99.2] | 97.0 [89.5 to 99.6]
  hSBA-MenC: >=1:4 | 98.7 [93.1 to 100.0] | 97.1 [90.1 to 99.7]
  hSBA-MenW-135: >=1:4: number analyzed (Participants) | 72 | 61
  hSBA-MenW-135: >=1:4 | 62.5 [50.3 to 73.6] | 68.9 [55.7 to 80.1]
  hSBA-MenY: >=1:4: number analyzed (Participants) | 71 | 56
  hSBA-MenY: >=1:4 | 67.6 [55.5 to 78.2] | 64.3 [50.4 to 76.6]
  hSBA-MenA: >=1:8: number analyzed (Participants) | 74 | 66
  hSBA-MenA: >=1:8 | 95.9 [88.6 to 99.2] | 97.0 [89.5 to 99.6]
  hSBA-MenC: >=1:8 | 98.7 [93.1 to 100.0] | 95.7 [88.0 to 99.1]
  hSBA-MenW-135: >=1:8: number analyzed (Participants) | 72 | 61
  hSBA-MenW-135: >=1:8 | 62.5 [50.3 to 73.6] | 68.9 [55.7 to 80.1]
  hSBA-MenY: >=1:8: number analyzed (Participants) | 71 | 56
  hSBA-MenY: >=1:8 | 67.6 [55.5 to 78.2] | 64.3 [50.4 to 76.6]

11. Secondary Outcome: Percentage of Participants With hSBA Titers >=1:4 and >=1:8 at 1 Month After Administration of 2 Doses of MenACWY-TT in the ACWY2d Group
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with hSBA titers >=1:4 and >=1:8 against each serogroup at 1 month after administration of 2 doses of MenACWY-TT are reported. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 2nd dose of MenACWY-TT (i.e. at Month 3)
Population: Analyzed on ATP cohort for persistence Year 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for ACWY1d, Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY2d Group
Number analyzed (Participants) | 70
percentage of participants
  hSBA-MenA: >=1:4: number analyzed (Participants) | 66
  hSBA-MenA: >=1:4 | 97.0 [89.5 to 99.6]
  hSBA-MenC: >=1:4: number analyzed (Participants) | 69
  hSBA-MenC: >=1:4 | 100.0 [94.8 to 100.0]
  hSBA-MenW-135: >=1:4 | 97.1 [90.1 to 99.7]
  hSBA-MenY: >=1:4: number analyzed (Participants) | 64
  hSBA-MenY: >=1:4 | 95.3 [86.9 to 99.0]
  hSBA-MenA: >=1:8: number analyzed (Participants) | 66
  hSBA-MenA: >=1:8 | 97.0 [89.5 to 99.6]
  hSBA-MenC: >=1:8: number analyzed (Participants) | 69
  hSBA-MenC: >=1:8 | 100.0 [94.8 to 100.0]
  hSBA-MenW-135: >=1:8 | 97.1 [90.1 to 99.7]
  hSBA-MenY: >=1:8: number analyzed (Participants) | 64
  hSBA-MenY: >=1:8 | 95.3 [86.9 to 99.0]

12. Secondary Outcome: Geometric Mean Titers (GMTs) With hSBA for Each of the 4 Serogroups Following Vaccination at 1 Month After Administration of 1 Dose of MenACWY-TT in the ACWY1d and ACWY2d Groups
Description: Geometric mean titers of antibodies against each serogroup were assessed using hSBA. Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). hSBA titers are expressed as 1/dilution. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 78 | 70
titers (1/dilution)
  hSBA-MenA: number analyzed (Participants) | 74 | 66
  hSBA-MenA | 118.0 [86.8 to 160.5] | 132.9 [98.1 to 180.1]
  hSBA-MenC | 151.9 [104.8 to 220.4] | 160.8 [109.8 to 235.5]
  hSBA-MenW-135: number analyzed (Participants) | 72 | 61
  hSBA-MenW-135 | 27.5 [16.1 to 46.8] | 26.2 [16.0 to 43.0]
  hSBA-MenY: number analyzed (Participants) | 71 | 56
  hSBA-MenY | 41.2 [23.7 to 71.5] | 31.9 [17.6 to 57.9]

13. Secondary Outcome: Geometric Mean Titers (GMTs) With hSBA for Each of the 4 Serogroups Following Vaccination at 1 Month After Administration of 2 Doses of MenACWY-TT in the ACWY2d Group
Description: as for outcome 12
Time Frame: 1 month after administration of 2nd dose of MenACWY-TT (i.e. at Month 3)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY2d Group
Number analyzed (Participants) | 70
titers (1/dilution)
  hSBA-MenA: number analyzed (Participants) | 66
  hSBA-MenA | 170.5 [126.2 to 230.2]
  hSBA-MenC: number analyzed (Participants) | 69
  hSBA-MenC | 1753.3 [1278.7 to 2404.2]
  hSBA-MenW-135 | 756.8 [550.1 to 1041.3]
  hSBA-MenY: number analyzed (Participants) | 64
  hSBA-MenY | 513.0 [339.4 to 775.4]

14. Secondary Outcome: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 at 1 Month After Administration of 1 Dose of MenACWY-TT in the PCV-13 Group
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 and >=1:128 against each serogroup at 1 month after administration of MenACWY-TT are reported. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 3)
Population: Analyzed on ATP cohort for persistence Year 1 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for ACWY1d, ACWY2d and Co-ad reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCV13 Group
Number analyzed (Participants) | 169
percentage of participants
  rSBA-MenA: >=1:8 | 96.4 [92.4 to 98.7]
  rSBA-MenC: >=1:8 | 95.3 [90.9 to 97.9]
  rSBA-MenW-135: >=1:8 | 96.4 [92.4 to 98.7]
  rSBA-MenY: >=1:8 | 97.0 [93.2 to 99.0]
  rSBA-MenA: >=1:128 | 95.9 [91.7 to 98.3]
  rSBA-MenC: >=1:128 | 85.8 [79.6 to 90.7]
  rSBA-MenW-135: >=1:128 | 96.4 [92.4 to 98.7]
  rSBA-MenY: >=1:128 | 97.0 [93.2 to 99.0]

15. Secondary Outcome: Geometric Mean Titers (GMTs) With rSBA Titers for Each of the 4 Serogroups Following Vaccination at 1 Month After Administration of 1 Dose of MenACWY-TT in the PCV-13 Group
Description: as for outcome 4
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 3)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | PCV13 Group
Number analyzed (Participants) | 169
titers (1/dilution)
  rSBA-MenA | 1957.7 [1513.4 to 2532.3]
  rSBA-MenC | 376.4 [284.7 to 497.6]
  rSBA-MenW-135 | 3490.5 [2643.3 to 4609.3]
  rSBA-MenY | 1481.2 [1158.4 to 1893.9]

16. Secondary Outcome: Percentage of Participants With rSBA Titers >=1:128 at 1 Month After Administration of 1 Dose of MenACWY-TT in the ACWY1d, ACWY2d and Co-ad Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:128 against each serogroup at 1 month after administration of MenACWY-TT are reported. ATP cohort for persistence Year 1 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group
Number analyzed (Participants) | 180 | 158 | 178
percentage of participants
  rSBA-MenA | 94.4 [90.0 to 97.3] | 95.6 [91.1 to 98.2] | 93.8 [89.2 to 96.9]
  rSBA-MenC: number analyzed (Participants) | 179 | 157 | 176
  rSBA-MenC | 85.5 [79.4 to 90.3] | 85.4 [78.8 to 90.5] | 88.1 [82.3 to 92.5]
  rSBA-MenW-135: number analyzed (Participants) | 180 | 158 | 177
  rSBA-MenW-135 | 95.0 [90.7 to 97.7] | 94.3 [89.5 to 97.4] | 92.7 [87.8 to 96.0]
  rSBA-MenY: number analyzed (Participants) | 180 | 157 | 177
  rSBA-MenY | 90.6 [85.3 to 94.4] | 91.7 [86.3 to 95.5] | 89.3 [83.7 to 93.4]

17. Secondary Outcome: Geometric Mean Titers (GMTs) With rSBA for Each of the 4 Serogroups Following Vaccination at 1 Month After Administration of 1 Dose of MenACWY-TT in ACWY1d, ACWY2d and Co-ad Groups
Description: as for outcome 4
Time Frame: 1 month after administration of 1st dose of MenACWY-TT (i.e. at Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group
Number analyzed (Participants) | 180 | 158 | 178
titers (1/dilution)
  rSBA-MenA | 1437.0 [1118.3 to 1846.6] | 1275.2 [970.5 to 1675.4] | 1146.4 [867.9 to 1514.3]
  rSBA-MenC: number analyzed (Participants) | 179 | 157 | 176
  rSBA-MenC | 452.3 [345.6 to 591.9] | 369.3 [280.9 to 485.5] | 337.3 [263.8 to 431.1]
  rSBA-MenW-135: number analyzed (Participants) | 180 | 158 | 177
  rSBA-MenW-135 | 2120.2 [1601.0 to 2807.8] | 2030.1 [1510.7 to 2728.2] | 1550.9 [1137.4 to 2114.7]
  rSBA-MenY: number analyzed (Participants) | 180 | 157 | 177
  rSBA-MenY | 951.8 [705.0 to 1284.9] | 933.3 [692.3 to 1258.3] | 778.5 [566.2 to 1070.4]

18. Secondary Outcome: Percentage of Participants With hSBA Titers >=1:4 and >=1:8 at Year 1, 3 and 5 in the ACWY1d and ACWY2d Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with hSBA titers >=1:4 and >=1:8 against each serogroup at Year 1, 3 and 5 after administration of MenACWY-TT are reported. ATP cohort for persistence Year 1, 3 and 5 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 1, Year 3, Year 5
Population: Analyzed on ATP cohort for persistence Year 1, 3 and 5 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Co-ad and PCV13 reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 72 | 65
percentage of participants
  hSBA-MenA: >=1:4 (Year 1): number analyzed (Participants) | 70 | 62
  hSBA-MenA: >=1:4 (Year 1) | 37.1 [25.9 to 49.5] | 35.5 [23.7 to 48.7]
  hSBA-MenC: >=1:4 (Year 1): number analyzed (Participants) | 71 | 63
  hSBA-MenC: >=1:4 (Year 1) | 81.7 [70.7 to 89.9] | 93.7 [84.5 to 98.2]
  hSBA-MenW-135: >=1:4 (Year 1) | 95.8 [88.3 to 99.1] | 98.5 [91.7 to 100.0]
  hSBA-MenY: >=1:4 (Year 1): number analyzed (Participants) | 62 | 58
  hSBA-MenY: >=1:4 (Year 1) | 91.9 [82.2 to 97.3] | 87.9 [76.7 to 95.0]
  hSBA-MenA: >=1:8 (Year 1): number analyzed (Participants) | 70 | 62
  hSBA-MenA: >=1:8 (Year 1) | 35.7 [24.6 to 48.1] | 35.5 [23.7 to 48.7]
  hSBA-MenC: >=1:8 (Year 1): number analyzed (Participants) | 71 | 63
  hSBA-MenC: >=1:8 (Year 1) | 80.3 [69.1 to 88.8] | 90.5 [80.4 to 96.4]
  hSBA-MenW-135: >=1:8 (Year 1) | 95.8 [88.3 to 99.1] | 98.5 [91.7 to 100.0]
  hSBA-MenY: >=1:8 (Year 1): number analyzed (Participants) | 62 | 58
  hSBA-MenY: >=1:8 (Year 1) | 91.9 [82.2 to 97.3] | 87.9 [76.7 to 95.0]
  hSBA-MenA: >=1:4 (Year 3): number analyzed (Participants) | 55 | 50
  hSBA-MenA: >=1:4 (Year 3) | 36.4 [23.8 to 50.4] | 36.0 [22.9 to 50.8]
  hSBA-MenC: >=1:4 (Year 3): number analyzed (Participants) | 61 | 56
  hSBA-MenC: >=1:4 (Year 3) | 65.6 [52.3 to 77.3] | 67.9 [54.0 to 79.7]
  hSBA-MenW-135: >=1:4 (Year 3): number analyzed (Participants) | 67 | 54
  hSBA-MenW-135: >=1:4 (Year 3) | 71.6 [59.3 to 82.0] | 87.0 [75.1 to 94.6]
  hSBA-MenY: >=1:4 (Year 3): number analyzed (Participants) | 64 | 52
  hSBA-MenY: >=1:4 (Year 3) | 53.1 [40.2 to 65.7] | 61.5 [47.0 to 74.7]
  hSBA-MenA: >=1:8 (Year 3): number analyzed (Participants) | 55 | 50
  hSBA-MenA: >=1:8 (Year 3) | 36.4 [23.8 to 50.4] | 36.0 [22.9 to 50.8]
  hSBA-MenC: >=1:8 (Year 3): number analyzed (Participants) | 61 | 56
  hSBA-MenC: >=1:8 (Year 3) | 65.6 [52.3 to 77.3] | 67.9 [54.0 to 79.7]
  hSBA-MenW-135: >=1:8 (Year 3): number analyzed (Participants) | 67 | 54
  hSBA-MenW-135: >=1:8 (Year 3) | 71.6 [59.3 to 82.0] | 87.0 [75.1 to 94.6]
  hSBA-MenY: >=1:8 (Year 3): number analyzed (Participants) | 64 | 52
  hSBA-MenY: >=1:8 (Year 3) | 53.1 [40.2 to 65.7] | 61.5 [47.0 to 74.7]
  hSBA-MenA: >=1:4 (Year 5): number analyzed (Participants) | 61 | 56
  hSBA-MenA: >=1:4 (Year 5) | 27.9 [17.1 to 40.8] | 17.9 [8.9 to 30.4]
  hSBA-MenC: >=1:4 (Year 5): number analyzed (Participants) | 61 | 59
  hSBA-MenC: >=1:4 (Year 5) | 60.7 [47.3 to 72.9] | 67.8 [54.4 to 79.4]
  hSBA-MenW-135: >=1:4 (Year 5): number analyzed (Participants) | 56 | 44
  hSBA-MenW-135: >=1:4 (Year 5) | 58.9 [45.0 to 71.9] | 63.6 [47.8 to 77.6]
  hSBA-MenY: >=1:4 (Year 5): number analyzed (Participants) | 65 | 48
  hSBA-MenY: >=1:4 (Year 5) | 61.5 [48.6 to 73.3] | 54.2 [39.2 to 68.6]
  hSBA-MenA: >=1:8 (Year 5): number analyzed (Participants) | 61 | 56
  hSBA-MenA: >=1:8 (Year 5) | 27.9 [17.1 to 40.8] | 17.9 [8.9 to 30.4]
  hSBA-MenC: >=1:8 (Year 5): number analyzed (Participants) | 61 | 59
  hSBA-MenC: >=1:8 (Year 5) | 60.7 [47.3 to 72.9] | 67.8 [54.4 to 79.4]
  hSBA-MenW-135: >=1:8 (Year 5): number analyzed (Participants) | 56 | 44
  hSBA-MenW-135: >=1:8 (Year 5) | 58.9 [45.0 to 71.9] | 63.6 [47.8 to 77.6]
  hSBA-MenY: >=1:8 (Year 5): number analyzed (Participants) | 65 | 48
  hSBA-MenY: >=1:8 (Year 5) | 61.5 [48.6 to 73.3] | 54.2 [39.2 to 68.6]

19. Secondary Outcome: Geometric Mean Titers (GMTs) With hSBA for Each of the 4 Serogroups Following Vaccination at Year 1, 3 and 5 in the ACWY1d and ACWY2d Groups
Description: Geometric mean titers of antibodies against each serogroup were assessed using hSBA. Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). hSBA titers are expressed as 1/dilution. ATP cohort for persistence Year 1, 3 and 5 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 1, Year 3, Year 5
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | ACWY1d Group | ACWY2d Group
Number analyzed (Participants) | 72 | 65
titers (1/dilution)
  hSBA-MenA (Year 1): number analyzed (Participants) | 70 | 62
  hSBA-MenA (Year 1) | 6.1 [4.1 to 8.9] | 6.4 [4.2 to 10.0]
  hSBA-MenC (Year 1): number analyzed (Participants) | 71 | 63
  hSBA-MenC (Year 1) | 35.2 [22.5 to 55.2] | 73.4 [47.5 to 113.4]
  hSBA-MenW-135 (Year 1) | 209.0 [149.9 to 291.4] | 232.6 [168.3 to 321.4]
  hSBA-MenY (Year 1): number analyzed (Participants) | 62 | 58
  hSBA-MenY (Year 1) | 144.4 [97.2 to 214.5] | 143.9 [88.5 to 233.8]
  hSBA-MenA (Year 3): number analyzed (Participants) | 55 | 50
  hSBA-MenA (Year 3) | 5.8 [3.8 to 8.9] | 5.4 [3.6 to 8.0]
  hSBA-MenC (Year 3): number analyzed (Participants) | 61 | 56
  hSBA-MenC (Year 3) | 23.6 [13.9 to 40.2] | 27.0 [15.6 to 46.8]
  hSBA-MenW-135 (Year 3): number analyzed (Participants) | 67 | 54
  hSBA-MenW-135 (Year 3) | 30.5 [18.7 to 49.6] | 55.5 [35.3 to 87.1]
  hSBA-MenY (Year 3): number analyzed (Participants) | 64 | 52
  hSBA-MenY (Year 3) | 17.3 [10.1 to 29.6] | 24.1 [13.3 to 43.8]
  hSBA-MenA (Year 5): number analyzed (Participants) | 61 | 56
  hSBA-MenA (Year 5) | 4.4 [3.1 to 6.2] | 3.1 [2.4 to 4.0]
  hSBA-MenC (Year 5): number analyzed (Participants) | 61 | 59
  hSBA-MenC (Year 5) | 18.1 [10.9 to 30.0] | 29.4 [16.3 to 52.9]
  hSBA-MenW-135 (Year 5): number analyzed (Participants) | 56 | 44
  hSBA-MenW-135 (Year 5) | 20.8 [11.6 to 37.1] | 19.5 [10.7 to 35.2]
  hSBA-MenY (Year 5): number analyzed (Participants) | 65 | 48
  hSBA-MenY (Year 5) | 24.3 [14.3 to 41.1] | 16.8 [9.0 to 31.3]

20. Secondary Outcome: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 at Year 1, 3 and 5 in the Co-ad and PCV-13 Groups
Description: Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). Percentage of participants with rSBA titers >=1:8 and >=1:128 against each serogroup at Year 1, 3 and 5 after administration of MenACWY-TT are reported. ATP cohort for persistence Year 1, 3 and 5 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 1, Year 3, Year 5
Population: Analyzed on ATP cohort for persistence Year 1, 3 and 5 population. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category. Data for this outcome measure was not planned to be collected and analyzed for ACWY1d and ACWY2d reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 173 | 169
percentage of participants
  rSBA-MenA: >=1:8 (Year 1) | 66.5 [58.9 to 73.5] | 70.4 [62.9 to 77.2]
  rSBA-MenC: >=1:8 (Year 1): number analyzed (Participants) | 171 | 169
  rSBA-MenC: >=1:8 (Year 1) | 42.7 [35.2 to 50.5] | 50.3 [42.5 to 58.1]
  rSBA-MenW-135: >=1:8 (Year 1): number analyzed (Participants) | 171 | 169
  rSBA-MenW-135: >=1:8 (Year 1) | 60.2 [52.5 to 67.6] | 72.8 [65.4 to 79.3]
  rSBA-MenY: >=1:8 (Year 1) | 67.1 [59.5 to 74.0] | 80.5 [73.7 to 86.2]
  rSBA-MenA: >=1:128 (Year 1) | 42.8 [35.3 to 50.5] | 56.2 [48.4 to 63.8]
  rSBA-MenC: >=1:128 (Year 1): number analyzed (Participants) | 171 | 169
  rSBA-MenC: >=1:128 (Year 1) | 15.8 [10.7 to 22.1] | 20.1 [14.4 to 27.0]
  rSBA-MenW-135: >=1:128 (Year 1): number analyzed (Participants) | 171 | 169
  rSBA-MenW-135: >=1:128 (Year 1) | 42.7 [35.2 to 50.5] | 58.0 [50.2 to 65.5]
  rSBA-MenY: >=1:128 (Year 1) | 53.8 [46.0 to 61.4] | 69.2 [61.7 to 76.1]
  rSBA-MenA: >=1:8 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenA: >=1:8 (Year 3) | 51.0 [42.7 to 59.2] | 53.8 [44.9 to 62.5]
  rSBA-MenC: >=1:8 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenC: >=1:8 (Year 3) | 28.5 [21.4 to 36.4] | 31.8 [24.0 to 40.5]
  rSBA-MenW-135: >=1:8 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenW-135: >=1:8 (Year 3) | 53.0 [44.7 to 61.1] | 56.8 [47.9 to 65.4]
  rSBA-MenY: >=1:8 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenY: >=1:8 (Year 3) | 62.9 [54.7 to 70.6] | 73.5 [65.1 to 80.8]
  rSBA-MenA: >=1:128 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenA: >=1:128 (Year 3) | 39.1 [31.2 to 47.3] | 40.2 [31.7 to 49.0]
  rSBA-MenC: >=1:128 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenC: >=1:128 (Year 3) | 14.6 [9.4 to 21.2] | 10.6 [5.9 to 17.2]
  rSBA-MenW-135: >=1:128 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenW-135: >=1:128 (Year 3) | 39.1 [31.2 to 47.3] | 42.4 [33.9 to 51.3]
  rSBA-MenY: >=1:128 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenY: >=1:128 (Year 3) | 53.0 [44.7 to 61.1] | 59.8 [51.0 to 68.3]
  rSBA-MenA: >=1:8 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenA: >=1:8 (Year 5) | 45.8 [37.4 to 54.3] | 47.3 [38.4 to 56.3]
  rSBA-MenC: >=1:8 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenC: >=1:8 (Year 5) | 23.9 [17.2 to 31.8] | 19.4 [13.0 to 27.3]
  rSBA-MenW-135: >=1:8 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenW-135: >=1:8 (Year 5) | 43.0 [34.7 to 51.5] | 45.0 [36.2 to 54.0]
  rSBA-MenY: >=1:8 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenY: >=1:8 (Year 5) | 52.8 [44.3 to 61.2] | 55.8 [46.8 to 64.5]
  rSBA-MenA: >=1:128 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenA: >=1:128 (Year 5) | 19.0 [12.9 to 26.4] | 36.4 [28.1 to 45.4]
  rSBA-MenC: >=1:128 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenC: >=1:128 (Year 5) | 12.0 [7.1 to 18.5] | 7.8 [3.8 to 13.8]
  rSBA-MenW-135: >=1:128 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenW-135: >=1:128 (Year 5) | 33.8 [26.1 to 42.2] | 35.7 [27.4 to 44.6]
  rSBA-MenY: >=1:128 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenY: >=1:128 (Year 5) | 42.3 [34.0 to 50.8] | 48.1 [39.2 to 57.0]

21. Secondary Outcome: Geometric Mean Titers (GMTs) With rSBA for Each of the 4 Serogroups Following Vaccination at Year 1, 3 and 5 in the Co-ad and PCV-13 Groups
Description: Geometric mean titers of antibodies against each serogroup were assessed using rSBA. Serogroups included neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY). rSBA titers are expressed as 1/dilution. ATP cohort for persistence Year 1, 3 and 5 included all participants who met eligibility criteria, received complete primary vaccination series, had assay results available for at least 1 antigen tested, complied with procedures and intervals in protocol, did not present medical condition, received product or were non-compliant with protocol-defined serum sampling windows or lack of availability of immunogenicity results at the previous time point.
Time Frame: At Year 1, Year 3, Year 5
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 173 | 169
titers (1/dilution)
  rSBA-MenA (Year 1) | 59.5 [40.7 to 87.2] | 119.4 [79.5 to 179.3]
  rSBA-MenC (Year 1): number analyzed (Participants) | 171 | 169
  rSBA-MenC (Year 1) | 12.6 [10.0 to 16.0] | 16.0 [12.2 to 20.9]
  rSBA-MenW-135 (Year 1): number analyzed (Participants) | 171 | 169
  rSBA-MenW-135 (Year 1) | 52.0 [35.5 to 76.4] | 109.5 [75.0 to 160.0]
  rSBA-MenY (Year 1) | 70.7 [49.0 to 102.1] | 169.2 [119.2 to 240.1]
  rSBA-MenA (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenA (Year 3) | 38.6 [25.4 to 58.8] | 42.3 [27.2 to 65.6]
  rSBA-MenC (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenC (Year 3) | 9.1 [7.1 to 11.6] | 9.3 [7.1 to 12.1]
  rSBA-MenW-135 (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenW-135 (Year 3) | 34.4 [23.4 to 50.6] | 44.5 [28.9 to 68.7]
  rSBA-MenY (Year 3): number analyzed (Participants) | 151 | 132
  rSBA-MenY (Year 3) | 67.6 [45.6 to 100.3] | 106.0 [70.2 to 160.0]
  rSBA-MenA (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenA (Year 5) | 15.4 [11.1 to 21.3] | 28.3 [18.5 to 43.2]
  rSBA-MenC (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenC (Year 5) | 7.9 [6.2 to 10.0] | 7.0 [5.5 to 8.8]
  rSBA-MenW-135 (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenW-135 (Year 5) | 26.2 [17.6 to 39.0] | 31.7 [20.2 to 49.6]
  rSBA-MenY (Year 5): number analyzed (Participants) | 142 | 129
  rSBA-MenY (Year 5) | 43.3 [28.3 to 66.2] | 53.9 [34.5 to 84.2]

22. Secondary Outcome: Percentage of Participants With Antibody Concentrations >=0.15 mcg/mL, >=0.26 mcg/mL and >=0.35 mcg/mL for Each of the Anti-pneumococcal Serotypes at 1 Month After Administration of Prevnar 13 in the Co-ad and PCV-13 Groups
Description: Antibody concentrations were determined for anti-pneumococcal antibodies: anti-1, anti-3, anti-4, anti-5, anti-6A, anti-6B, anti-7F, anti-9V, anti-14, anti-18C, anti-19A, anti-19F and anti-23F. Percentage of participants with antibody concentrations >=0.15 mcg/mL, >=0.26 mcg/mL and >=0.35 mcg/mL against each serogroup at 1 month after administration of Prevnar 13 are reported. ATP cohort for immunogenicity post dose 1 included all evaluable participants who met eligibility criteria, complied with the procedures defined in the protocol and with no elimination criteria during the study from the ATP cohort for safety, received all study vaccines at Month 0, had assay results available for antibodies against at least one study vaccine antigen component at Visit 2, those with available blood sample at Visit 2 for PCV13 group.
Time Frame: 1 month after administration of Prevnar 13 (i.e. at Month 1)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 163 | 172
percentage of participants
  anti-1 (>=0.15 mcg/mL): number analyzed (Participants) | 162 | 171
  anti-1 (>=0.15 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-3 (>=0.15 mcg/mL): number analyzed (Participants) | 151 | 162
  anti-3 (>=0.15 mcg/mL) | 99.3 [96.4 to 100] | 97.5 [93.8 to 99.3]
  anti-4 (>=0.15 mcg/mL) | 100 [97.8 to 100] | 99.4 [96.8 to 100]
  anti-5 (>=0.15 mcg/mL) | 100 [97.8 to 100] | 100 [97.9 to 100]
  anti-6A (>=0.15 mcg/mL): number analyzed (Participants) | 163 | 171
  anti-6A (>=0.15 mcg/mL) | 100 [97.8 to 100] | 100 [97.9 to 100]
  anti-6B (>=0.15 mcg/mL): number analyzed (Participants) | 161 | 171
  anti-6B (>=0.15 mcg/mL) | 100 [97.7 to 100] | 99.4 [96.8 to 100]
  anti-7F (>=0.15 mcg/mL) | 100 [97.8 to 100] | 100 [97.9 to 100]
  anti-9V (>=0.15 mcg/mL) | 99.4 [96.6 to 100] | 100 [97.9 to 100]
  anti-14 (>=0.15 mcg/mL): number analyzed (Participants) | 161 | 172
  anti-14 (>=0.15 mcg/mL) | 100 [97.7 to 100] | 99.4 [96.8 to 100]
  anti-18C (>=0.15 mcg/mL) | 100 [97.8 to 100] | 100 [97.9 to 100]
  anti-19A (>=0.15 mcg/mL): number analyzed (Participants) | 162 | 170
  anti-19A (>=0.15 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-19F (>=0.15 mcg/mL): number analyzed (Participants) | 162 | 172
  anti-19F (>=0.15 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-23F (>=0.15 mcg/mL): number analyzed (Participants) | 161 | 169
  anti-23F (>=0.15 mcg/mL) | 100 [97.7 to 100] | 100 [97.8 to 100]
  anti-1 (>=0.26 mcg/mL): number analyzed (Participants) | 162 | 171
  anti-1 (>=0.26 mcg/mL) | 99.4 [96.6 to 100] | 99.4 [96.8 to 100]
  anti-3 (>=0.26 mcg/mL): number analyzed (Participants) | 151 | 162
  anti-3 (>=0.26 mcg/mL) | 94.0 [89.0 to 97.2] | 88.3 [82.3 to 92.8]
  anti-4 (>=0.26 mcg/mL) | 98.8 [95.6 to 99.9] | 98.3 [95.0 to 99.6]
  anti-5 (>=0.26 mcg/mL) | 99.4 [96.6 to 100] | 98.8 [95.9 to 99.9]
  anti-6A (>=0.26 mcg/mL): number analyzed (Participants) | 163 | 171
  anti-6A (>=0.26 mcg/mL) | 100 [97.8 to 100] | 100 [97.9 to 100]
  anti-6B (>=0.26 mcg/mL): number analyzed (Participants) | 161 | 171
  anti-6B (>=0.26 mcg/mL) | 100 [97.7 to 100] | 99.4 [96.8 to 100]
  anti-7F (>=0.26 mcg/mL) | 100 [97.8 to 100] | 100 [97.9 to 100]
  anti-9V (>=0.26 mcg/mL) | 99.4 [96.6 to 100] | 98.8 [95.9 to 99.9]
  anti-14 (>=0.26 mcg/mL): number analyzed (Participants) | 161 | 172
  anti-14 (>=0.26 mcg/mL) | 100 [97.7 to 100] | 99.4 [96.8 to 100]
  anti-18C (>=0.26 mcg/mL) | 98.8 [95.6 to 99.9] | 99.4 [96.8 to 100]
  anti-19A (>=0.26 mcg/mL): number analyzed (Participants) | 162 | 170
  anti-19A (>=0.26 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-19F (>=0.26 mcg/mL): number analyzed (Participants) | 162 | 172
  anti-19F (>=0.26 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-23F (>=0.26 mcg/mL): number analyzed (Participants) | 161 | 169
  anti-23F (>=0.26 mcg/mL) | 99.4 [96.6 to 100] | 99.4 [96.7 to 100]
  anti-1 (>=0.35 mcg/mL): number analyzed (Participants) | 162 | 171
  anti-1 (>=0.35 mcg/mL) | 99.4 [96.6 to 100] | 98.2 [95.0 to 99.6]
  anti-3 (>=0.35 mcg/mL): number analyzed (Participants) | 151 | 162
  anti-3 (>=0.35 mcg/mL) | 83.4 [76.5 to 89.0] | 79.0 [71.9 to 85.0]
  anti-4 (>=0.35 mcg/mL) | 96.9 [93.0 to 99.0] | 97.1 [93.3 to 99.0]
  anti-5 (>=0.35 mcg/mL) | 98.8 [95.6 to 99.9] | 94.8 [90.3 to 97.6]
  anti-6A (>=0.35 mcg/mL): number analyzed (Participants) | 163 | 171
  anti-6A (>=0.35 mcg/mL) | 99.4 [96.6 to 100] | 100 [97.9 to 100]
  anti-6B (>=0.35 mcg/mL): number analyzed (Participants) | 161 | 171
  anti-6B (>=0.35 mcg/mL) | 99.4 [96.6 to 100] | 99.4 [96.8 to 100]
  anti-7F (>=0.35 mcg/mL) | 99.4 [96.6 to 100] | 100 [97.9 to 100]
  anti-9V (>=0.35 mcg/mL) | 99.4 [96.6 to 100] | 97.7 [94.2 to 99.4]
  anti-14 (>=0.35 mcg/mL): number analyzed (Participants) | 161 | 172
  anti-14 (>=0.35 mcg/mL) | 100 [97.7 to 100] | 99.4 [96.8 to 100]
  anti-18C (>=0.35 mcg/mL) | 98.8 [95.6 to 99.9] | 99.4 [96.8 to 100]
  anti-19A (>=0.35 mcg/mL): number analyzed (Participants) | 162 | 170
  anti-19A (>=0.35 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-19F (>=0.35 mcg/mL): number analyzed (Participants) | 162 | 172
  anti-19F (>=0.35 mcg/mL) | 100 [97.7 to 100] | 100 [97.9 to 100]
  anti-23F (>=0.35 mcg/mL): number analyzed (Participants) | 161 | 169
  anti-23F (>=0.35 mcg/mL) | 99.4 [96.6 to 100] | 99.4 [96.7 to 100]

23. Secondary Outcome: Percentage of Participants With Opsonophagocytic Activity (OPA) Titers >=1:8 for Each of the Anti-pneumococcal Serotypes at 1 Month After Administration of Prevnar 13 in the Co-ad and PCV-13 Groups
Description: OPA titers were determined for anti-pneumococcal serotypes: OPSONO-1, OPSONO-3, OPSONO-4, OPSONO-5, OPSONO-6A, OPSONO-6B, OPSONO-7F, OPSONO-9V, OPSONO-14, OPSONO-18C, OPSONO-19A, OPSONO-19F and OPSONO-23F. Percentage of participants with OPA titers >=1:8 against each serogroup at 1 month after administration of Prevnar 13 are reported. ATP cohort for immunogenicity post dose 1 included all evaluable participants who met eligibility criteria, complied with the procedures defined in the protocol and with no elimination criteria during the study from the ATP cohort for safety, received all study vaccines at Month 0, had assay results available for antibodies against at least one study vaccine antigen component at Visit 2, those with available blood sample at Visit 2 for PCV13 group.
Time Frame: 1 month after administration of Prevnar 13 (i.e. at Month 1)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 81 | 88
percentage of participants
  OPSONO-1: number analyzed (Participants) | 81 | 86
  OPSONO-1 | 93.8 [86.2 to 98.0] | 90.7 [82.5 to 95.9]
  OPSONO-3: number analyzed (Participants) | 76 | 80
  OPSONO-3 | 98.7 [92.9 to 100] | 100 [95.5 to 100]
  OPSONO-4: number analyzed (Participants) | 77 | 80
  OPSONO-4 | 100 [95.3 to 100] | 100 [95.5 to 100]
  OPSONO-5: number analyzed (Participants) | 81 | 87
  OPSONO-5 | 100 [95.5 to 100] | 100 [95.8 to 100]
  OPSONO-6A | 100 [95.5 to 100] | 100 [95.9 to 100]
  OPSONO-6B: number analyzed (Participants) | 75 | 78
  OPSONO-6B | 100 [95.2 to 100] | 100 [95.4 to 100]
  OPSONO-7F: number analyzed (Participants) | 81 | 87
  OPSONO-7F | 100 [95.5 to 100] | 100 [95.8 to 100]
  OPSONO-9V | 100 [95.5 to 100] | 100 [95.9 to 100]
  OPSONO-14: number analyzed (Participants) | 73 | 78
  OPSONO-14 | 100 [95.1 to 100] | 100 [95.4 to 100]
  OPSONO-18C | 100 [95.5 to 100] | 100 [95.9 to 100]
  OPSONO-19A | 100 [95.5 to 100] | 100 [95.9 to 100]
  OPSONO-19F | 98.8 [93.3 to 100] | 100 [95.9 to 100]
  OPSONO-23F: number analyzed (Participants) | 77 | 80
  OPSONO-23F | 98.7 [93.0 to 100] | 98.8 [93.2 to 100]

24. Secondary Outcome: Geometric Mean Titers (GMTs) With OPA for Each of the Anti-pneumococcal Serotypes at 1 Month After Administration of Prevnar 13 in the Co-ad and PCV-13 Groups
Description: OPA titers were determined for anti-pneumococcal serotypes: OPSONO-1, OPSONO-3, OPSONO-4, OPSONO-5, OPSONO-6A, OPSONO-6B, OPSONO-7F, OPSONO-9V, OPSONO-14, OPSONO-18C, OPSONO-19A, OPSONO-19F and OPSONO-23F. OPA titers are expressed as 1/dilution. ATP cohort for immunogenicity post dose 1 included all evaluable participants who met eligibility criteria, complied with the procedures defined in the protocol and with no elimination criteria during the study from the ATP cohort for safety, received all study vaccines at Month 0, had assay results available for antibodies against at least one study vaccine antigen component at Visit 2, those with available blood sample at Visit 2 for PCV13 group.
Time Frame: 1 month after administration of Prevnar 13 (i.e. at Month 1)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 81 | 88
titers
  OPSONO-1: number analyzed (Participants) | 81 | 86
  OPSONO-1 | 116.1 [83.8 to 160.7] | 106.1 [77.0 to 146.2]
  OPSONO-3: number analyzed (Participants) | 76 | 80
  OPSONO-3 | 137.6 [106.4 to 178.0] | 122.0 [100.6 to 147.9]
  OPSONO-4: number analyzed (Participants) | 77 | 80
  OPSONO-4 | 2194.8 [1660.0 to 2901.9] | 2210.1 [1735.0 to 2815.2]
  OPSONO-5: number analyzed (Participants) | 81 | 87
  OPSONO-5 | 452.3 [360.4 to 567.5] | 404.6 [319.1 to 512.9]
  OPSONO-6A | 10177.2 [7784.7 to 13305.1] | 7354.2 [5707.4 to 9476.1]
  OPSONO-6B: number analyzed (Participants) | 75 | 78
  OPSONO-6B | 4952.3 [3734.4 to 6567.4] | 3881.5 [3055.8 to 4930.2]
  OPSONO-7F: number analyzed (Participants) | 81 | 87
  OPSONO-7F | 8957.4 [7306.4 to 10981.5] | 8526.5 [6926.2 to 10496.7]
  OPSONO-9V | 3375.5 [2539.6 to 4486.6] | 2332.3 [1766.1 to 3080.1]
  OPSONO-14: number analyzed (Participants) | 73 | 78
  OPSONO-14 | 3443.7 [2453.5 to 4833.5] | 3157.8 [2445.4 to 4077.8]
  OPSONO-18C | 3881.0 [2947.2 to 5110.7] | 3289.8 [2513.7 to 4305.5]
  OPSONO-19A | 3362.5 [2639.6 to 4283.4] | 2494.3 [1986.7 to 3131.6]
  OPSONO-19F | 1795.5 [1305.6 to 2469.2] | 1647.6 [1287.6 to 2108.3]
  OPSONO-23F: number analyzed (Participants) | 77 | 80
  OPSONO-23F | 7755.7 [5450.9 to 11034.9] | 5677.4 [4255.0 to 7575.3]

25. Secondary Outcome: Number of Participants With Solicited Local Reactions Within 4 Days Post Each Vaccination
Description: Solicited local reactions included pain, redness and swelling. Here, '0' in the number analyzed field signifies that no vaccine was administered in the specified group for the specified category.
Time Frame: Within 4 days post each vaccination (vaccination 1 [at Month 0] and vaccination 2 [at Month 2])
Population: The total vaccinated cohort (TVC) included all participants vaccinated with at least 1 dose of study vaccine. The analysis was performed per vaccine actually administered at Dose 1. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 199 | 196 | 197 | 197
Participants
  Pain: Post MenACWY-TT Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 0
  Pain: Post MenACWY-TT Dose 1 | 52 | 64 | 72 |
  Pain: Post Prevenar 13 Dose 1: number analyzed (Participants) | 0 | 0 | 196 | 196
  Pain: Post Prevenar 13 Dose 1 |  |  | 85 | 72
  Pain: Post MenACWY-TT Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Pain: Post MenACWY-TT Dose 2 |  | 58 |  | 53
  Redness: Post MenACWY-TT Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 0
  Redness: Post MenACWY-TT Dose 1 | 68 | 73 | 73 |
  Redness: Post Prevenar 13 Dose 1: number analyzed (Participants) | 0 | 0 | 196 | 196
  Redness: Post Prevenar 13 Dose 1 |  |  | 87 | 90
  Redness: Post MenACWY-TT Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Redness: Post MenACWY-TT Dose 2 |  | 64 |  | 66
  Swelling: Post MenACWY-TT Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 0
  Swelling: Post MenACWY-TT Dose 1 | 35 | 45 | 43 |
  Swelling: Post Prevenar 13 Dose 1: number analyzed (Participants) | 0 | 0 | 196 | 196
  Swelling: Post Prevenar 13 Dose 1 |  |  | 69 | 63
  Swelling: Post MenACWY-TT Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Swelling: Post MenACWY-TT Dose 2 |  | 34 |  | 30

26. Secondary Outcome: Number of Participants With Solicited General Reactions Within 4 Days Post Each Vaccination
Description: Solicited general reactions included drowsiness, irritability/fussiness, loss of appetite and fever. Here, '0' in the number analyzed field signifies that no vaccine was administered in the specified group for the specified category. Post dose 1 for ACWY1d and Co-ad group included reactions occurred after dosing of both MenACWY-TT and Prevenar 13 for Co-ad group and data was collected and summarized collectively.
Time Frame: Within 4 days post each vaccination (vaccination 1 [Dose 1] and vaccination 2 [Dose 2])
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 199 | 196 | 197 | 197
Participants
  Drowsiness: Post Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 196
  Drowsiness: Post Dose 1 | 62 | 73 | 85 | 72
  Drowsiness: Post Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Drowsiness: Post Dose 2 |  | 60 |  | 50
  Irritability/Fussiness: Post Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 196
  Irritability/Fussiness: Post Dose 1 | 89 | 93 | 107 | 85
  Irritability/Fussiness: Post Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Irritability/Fussiness: Post Dose 2 |  | 76 |  | 67
  Loss of Appetite: Post Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 196
  Loss of Appetite: Post Dose 1 | 56 | 60 | 54 | 58
  Loss of Appetite: Post Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Loss of Appetite: Post Dose 2 |  | 45 |  | 47
  Fever: Post Dose 1: number analyzed (Participants) | 199 | 195 | 197 | 196
  Fever: Post Dose 1 | 26 | 25 | 34 | 43
  Fever: Post Dose 2: number analyzed (Participants) | 0 | 189 | 0 | 191
  Fever: Post Dose 2 |  | 23 |  | 25

27. Secondary Outcome: Number of Participants With Unsolicited Adverse Events Within 31 Days Post Any Study Vaccination, Classified According to Medical Dictionary for Regulatory Activities (MedDRA)
Description: An adverse event was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited adverse event was an observed adverse event that did not fulfill the conditions prelisted in the case report book (CRB) in terms of symptom and/or onset post-vaccination.
Time Frame: Within 31 days post any vaccination
Population: The total vaccinated cohort (TVC) included all participants vaccinated with at least 1 dose of study vaccine. The analysis was performed per vaccine actually administered at Dose 1.
Measure: Count of Participants; unit: Participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 203 | 197 | 201 | 201
Participants | 11 | 15 | 11 | 11

28. Secondary Outcome: Number of Participants With Serious Adverse Events From Month 0 to Month 9
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect.
Time Frame: Month 0 to Month 9
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 203 | 197 | 201 | 201
Participants | 8 | 6 | 10 | 5

29. Secondary Outcome: Number of Participants With Serious Adverse Events Related to Study Vaccination From First Dose of Study Drug up to End of Study
Description: An adverse event was any untoward medical occurrence in a participant who received study drug. Serious adverse event was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Related adverse events were those adverse events who were related to the vaccination as judged by the investigator.
Time Frame: Baseline up to end of study (up to 5 years)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 203 | 197 | 201 | 201
Participants | 0 | 2 | 1 | 0

30. Secondary Outcome: Number of Participants With Any New Onset of Chronic Illnesses (NOCIs) From Month 0 to Month 9
Description: New onset chronic illness included autoimmune disorders, asthma, type I diabetes and allergies.
Time Frame: Month 0 to Month 9
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
Number analyzed (Participants) | 203 | 197 | 201 | 201
Participants | 2 | 3 | 1 | 5

ADVERSE EVENTS:
Time Frame: AE data were collected from Baseline up to end of study (up to 5 years). Solicited local and general reactions was collected within 4 days post vaccination.
Description: Same event may appear as both an adverse event and serious adverse events. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | ACWY1d Group | ACWY2d Group | Co-ad Group | PCV13 Group
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/197 | 1/201 | 1/201
Serious Adverse Events (participants affected / at risk) | 12/203 | 11/197 | 13/201 | 16/201
Other Adverse Events (participants affected / at risk) | 199/203 | 196/197 | 197/201 | 197/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACWY1d Group (N=203) | ACWY2d Group (N=197) | Co-ad Group (N=201) | PCV13 Group (N=201)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 1
Myringitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3 | 3 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Petroleum distillate poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ACWY1d Group (N=203) | ACWY2d Group (N=197) | Co-ad Group (N=201) | PCV13 Group (N=201)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 14 | 9 | 23
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Teething (Gastrointestinal disorders) | 7 | 14 | 12 | 18
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 17 | 4 | 7
Crying (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 2
Injection site bruising (General disorders) | 1 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 12 | 19 | 12 | 13
Swelling face (General disorders) | 0 | 1 | 0 | 0
Vaccination site bruising (General disorders) | 1 | 1 | 1 | 2
Vaccination site pain (General disorders) | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 3 | 2 | 7
Bronchitis (Infections and infestations) | 2 | 3 | 1 | 4
Conjunctivitis (Infections and infestations) | 2 | 9 | 4 | 9
Coxsackie viral infection (Infections and infestations) | 1 | 2 | 0 | 1
Croup infectious (Infections and infestations) | 0 | 3 | 2 | 3
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 6 | 1 | 3
Erythema infectiosum (Infections and infestations) | 1 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 2
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 2 | 6
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 4 | 6 | 4
Herpangina (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 2 | 0 | 1
Infected bite (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 4 | 2
Laryngitis (Infections and infestations) | 1 | 1 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Measles (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 17 | 11 | 15
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 3 | 8 | 4 | 11
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Otosalpingitis (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 3 | 2 | 2
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 4 | 5 | 3 | 4
Roseola (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 5 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 12 | 28 | 15 | 24
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 2 | 4 | 1 | 2
Viral infection (Infections and infestations) | 6 | 12 | 4 | 7
Viral rash (Infections and infestations) | 1 | 2 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 4 | 1 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Body temperature (Investigations) | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 3 | 1 | 0 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Autism spectrum disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Fear (Psychiatric disorders) | 1 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 6 | 5 | 3
Sleep disorder (Psychiatric disorders) | 0 | 3 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Genital labial adhesions (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal adhesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 21 | 8 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 6
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal mucosal discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 6 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 5
Eczema (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 5
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 9 | 5 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 52/199 | 91/196 | 94/197 | 91/197 — Number of participants evaluable for this local reaction.
Redness (General disorders) | 68/199 | 88/196 | 94/197 | 108/197 — Number of participants evaluable for this local reaction.
Swelling (General disorders) | 35/199 | 57/196 | 75/197 | 73/197 — Number of participants evaluable for this local reaction.
Drowsiness (General disorders) | 62/199 | 99/196 | 85/197 | 89/197 — Number of participants evaluable for this general reaction.
Irritability/Fussiness (General disorders) | 89/199 | 116/196 | 107/197 | 108/197 — Number of participants evaluable for this general reaction.
Loss Of Appetite (General disorders) | 56/199 | 78/196 | 54/197 | 83/197 — Number of participants evaluable for this general reaction.
Temperature/(Rectal) (°C) (General disorders) | 26/199 | 46/196 | 34/197 | 63/197 — Number of participants evaluable for this general reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT01939158/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT01939158/SAP_001.pdf